CLINICAL TRIAL: NCT05943535
Title: A Randomized, Double-blind, Placebo-controlled, Multinational, Phase 3 Study of the Efficacy and Safety of Inhaled Treprostinil in Subjects With Progressive Pulmonary Fibrosis (TETON-PPF)
Brief Title: Study of the Efficacy and Safety of Inhaled Treprostinil in Subjects With Progressive Pulmonary Fibrosis (TETON-PPF)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN-PF-305
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Progressive Pulmonary Fibrosis; Interstitial Lung Disease
Keywords: Treprostinil; PPF; ILD
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo inhaled using an ultrasonic nebulizer QID
  Interventions: Drug: Placebo; Device: Treprostinil Ultrasonic Nebulizer
- Inhaled Treprostinil (Experimental): Treprostinil for inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath. Inhaled QID and titrated up to a target of 12 breaths QID or until the subject reaches their maximum clinically tolerated dose.
  Interventions: Drug: Inhaled Treprostinil; Device: Treprostinil Ultrasonic Nebulizer

INTERVENTIONS:
Drug: Placebo — Placebo administered QID
  Arms: Placebo
Drug: Inhaled Treprostinil — Inhaled treprostinil (6 mcg/breath) administered QID
  Other Names: Tyvaso
  Arms: Inhaled Treprostinil
Device: Treprostinil Ultrasonic Nebulizer — Treprostinil ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath.

SUMMARY:
Study RIN-PF-305 is designed to evaluate the safety and efficacy of inhaled treprostinil in subjects with progressive pulmonary fibrosis (PPF) over a 52-week period.

DETAILED DESCRIPTION:
Study RIN-PF-305 is a Phase 3, multinational, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of inhaled treprostinil in subjects with PPF over a 52-week period. Subjects will be randomly allocated 1:1 to receive inhaled treprostinil or placebo. All subjects will initiate inhaled treprostinil or placebo at a dose of 3 breaths administered 4 times daily (QID) and will titrate to a target dosing regimen of 12 breaths QID. Study drug doses may be titrated up as tolerated, until the target dose or maximum clinically tolerated dose is achieved. Once eligible, 6 Treatment Period visits to the clinic will be required at Weeks 4, 8, 16, 28, 40, and 52.

Efficacy assessments include spirometry (forced vital capacity [FVC]), time to clinical worsening, time to first acute exacerbation of interstitial lung disease (ILD), overall survival, King's Brief Interstitial Lung Disease (K-BILD) questionnaire, plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) concentration, supplemental oxygen use, and lung diffusion capacity (DLCO). Safety assessments include the development of adverse events (AEs)/serious adverse events (SAEs), vital signs, clinical laboratory parameters, and electrocardiogram (ECG) parameters.

Subjects who complete the Week 52 Visit may be offered the opportunity to enter an open-label extension (OLE) study after completing the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject gives voluntary informed consent to participate in the study.
2. Subject is ≥18 years of age, inclusive, at the time of signing informed consent.
3. Subject has radiological evidence of pulmonary fibrosis of >10% extent on an HRCT scan in the previous 12 months (confirmed by central review).
4. Subject has a diagnosis of PPF (other than IPF) that fulfills at least 1 of the following criteria for progression within 24 months of screening despite standard treatment of ILD, as assessed by the Investigator:

   1. Clinically significant decline in % predicted FVC based on ≥10% relative decline
   2. Marginal decline in % predicted FVC based on ≥5% to <10% relative decline combined with worsening of respiratory symptoms
   3. Marginal decline in % predicted FVC based on ≥5% to <10% relative decline combined with increasing extent of fibrotic changes on chest imaging
   4. Worsening of respiratory symptoms as well as increasing extent of fibrotic changes on chest imaging
5. FVC ≥45% predicted at Screening (confirmed by central review).
6. Subjects must be on 1 of the following:

   1. On nintedanib or pirfenidone for ≥90 days prior to Baseline and in the Investigator's opinion, are planning to continue treatment through the study
   2. Not on treatment with nintedanib or pirfenidone for ≥90 days prior to Baseline and in the Investigator's opinion, not planning to initiate either treatment during the study.

   Concomitant use of both nintedanib and pirfenidone is not permitted.
7. Subjects treated with immunosuppressive agents (eg, mycophenolate, methotrexate, azathioprine, oral corticosteroids, rituximab) need to be on treatment for at least 120 days prior to Baseline and, in the Investigator's clinical opinion, must be refractory to treatment.
8. Women of childbearing potential must be non-pregnant (as confirmed by a urine pregnancy test at Screening and Baseline) and non-lactating, and will agree to do 1 of the following:

   1. Abstain from intercourse (when it is in line with their preferred and usual lifestyle)
   2. Use 2 medically acceptable, highly effective forms of contraception for the duration of the study, and at least 30 days after discontinuing study drug.

   i. Medically acceptable, highly effective forms of contraception can include approved hormonal contraceptives (oral, injectable, and implantable) and barrier methods (such as a condom or diaphragm) when used with a spermicide.

   Women who are successfully sterilized (including hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal (defined as amenorrhea for at least 12 consecutive months) are not considered to be of reproductive potential.
9. Males with a partner of childbearing potential must agree to use a condom for the duration of treatment and for at least 48 hours after discontinuing study drug.
10. In the opinion of the Investigator, the subject is able to communicate effectively with study personnel, and is considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

1. Subject is pregnant or lactating.
2. Subject has primary obstructive airway physiology (forced expiratory volume in 1 second/FVC <0.70 at Screening) or greater extent of emphysema than fibrosis on HRCT (confirmed by central review).
3. Subject has a diagnosis of IPF.
4. Subject has shown intolerance or significant lack of efficacy to a prostacyclin or prostacyclin analogue that resulted in discontinuation or inability to effectively titrate that therapy.
5. Subject has received any PAH-approved therapy, including prostacyclin therapy (epoprostenol, treprostinil, iloprost, or beraprost; except for acute vasoreactivity testing), IP receptor agonists (selexipag), endothelin receptor antagonists, phosphodiesterase type 5 inhibitors (PDE5-Is), soluble guanylate cyclase stimulators, or activin signaling inhibitors (sotatercept) within 60 days prior to Baseline. As needed use of a PDE5-I for erectile dysfunction is permitted, provided no doses are taken within 48 hours prior to any study-related efficacy assessments.
6. Subject is receiving >10 L/min of oxygen supplementation by any mode of delivery at rest at Baseline.
7. Exacerbation of ILD or active pulmonary or upper respiratory infection within 30 days prior to Baseline. Subjects must have completed any antibiotic or steroid regimens for treatment of the infection or acute exacerbation more than 30 days prior to Baseline to be eligible. If hospitalized for an acute exacerbation of ILD or a pulmonary or upper respiratory infection, subjects must have been discharged more than 90 days prior to Baseline to be eligible.
8. Subject has uncontrolled cardiac disease, defined as myocardial infarction within 6 months prior to Baseline or unstable angina within 30 days prior to Baseline.
9. Use of any other investigational drug/device or participation in any investigational study in which the subject received a medical intervention (ie, procedure, device, medication/supplement) within 30 days prior to Screening. Subjects participating in non-interventional, observational, or registry studies are eligible.
10. Acute pulmonary embolism within 90 days prior to Baseline.
11. In the opinion of the Investigator, the subject has any condition that would interfere with the interpretation of study assessments or would impair study participation or cooperation.
12. In the opinion of the Investigator, life expectancy <12 months due to ILD or a concomitant illness.
13. Subject has received nerandomilast within 60 days prior to Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Absolute FVC from Baseline to Week 52 | Baseline to Week 52
  The FVC measurement indicates the amount of air a person can forcefully and quickly exhale after taking a deep breath.

SECONDARY OUTCOMES:
Time to First Clinical Worsening | Baseline to Week 52
  Clinical worsening is monitored from randomization until 1 of the following criteria are met: death (all causes), hospitalization due to a respiratory indication, or ≥10% relative decline in % predicted FVC.
Time to First Acute Exacerbation of ILD | Baseline to Week 52
  An exacerbation of ILD is defined as an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality.
Overall Survival at Week 52 | Week 52
  Vital status will be assessed for all subjects at Week 52, including those who discontinue the study prematurely or who withdraw consent.
Change in % Predicted FVC from Baseline to Week 52 | Baseline to Week 52
  The FVC measurement indicates the amount of air a person can forcefully and quickly exhale after taking a deep breath. Percent predicted FVC is calculated based on factors such as race, sex, age, height, and weight.
Change in K-BILD Questionnaire Score from Baseline to Week 52 | Baseline to Week 52
  The K-BILD is a self-administered, 15-item questionnaire validated for patients with ILD consisting of 3 domains (breathlessness and activities, psychological, and chest symptoms).
Change in DLCO from Baseline to Week 52 | Baseline to Week 52
  The DLCO measurement measures how well oxygen moves from the lungs to the blood.

CONTACTS AND LOCATIONS:
Locations (148):
- United States (66):
  - UAB Lung Health Center, Birmingham, Alabama
  - Banner University Medical Center Phoenix Lung Institute, Phoenix, Arizona
  - Norton Thoracic Institute, Phoenix, Arizona
  - Peter Morton Medical Building, Los Angeles, California
  - NewportNativeMD, Inc., Newport Beach, California
  - University of California Irvine Medical Center, Orange, California
  - Paradigm Clinical Research, Redding, California
  - UC Davis Health Medical Center, Sacramento, California
  - Paradigm Clinical Research, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Ascension Medical Group St. Vincent's Lung Institute, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - TGH/USF Center for Advanced Lung Disease and Lung Transplant, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern Memorial Hospital, Clinical Research Unit, Chicago, Illinois
  - Rush University Medical Center Outpatient Pulmonary Clinic, Chicago, Illinois
  - UI Health Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville Healthcare Outpatient Research Clinic, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Adventist Healthcare White Oak Medical Center, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Infinity Medical Center, North Dartmouth, Massachusetts
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - University of Minnesota Health Clinical Research Unit (CRU), Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Northwell Health, New Hyde Park, New York
  - Weill Cornell Medicine, New York-Presbyterian Hospital, New York, New York
  - Stony Brook Advanced Specialty Care, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - PulmonIx LLC, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical CEnter, Columbus, Ohio
  - Mercy Health St.Vincent Medical Center LLC, Toledo, Ohio
  - Pennsylvania State Hershey Medical Center and College of Medicine, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina-Nexus, Charleston, South Carolina
  - Prisma Health Pulmonology-Richland, Columbia, South Carolina
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - StatCare Pulmonary Consultants, PLLC, Knoxville, Tennessee
  - The Vanderbilt Lung Institute, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center-Advanced Lung Clinic, Dallas, Texas
  - Houston Methodist Outpatient Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, McGovern Medical School, Houston, Texas
  - A & A Research Consultants, LLC, McAllen, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Christopher King, MD, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - University Hospital and UW Health Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (9):
  - Instituto Ave Pulmo - Fundacion enfisema, Mar del Plata, Buenos Aires
  - Instituto Medico Rio Cuarto, Río Cuarto, Córdoba Province
  - Sanatorio Parque de Rosario - Consultorios Externos, Rosario, Santa Fe Province
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
  - CIMER-Centro Integral de Medicina Respiratoria, San Miguel de Tucumán, Tucumán Province
  - CINME Centro de Investigaciones Metabolicas, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Instituto de Medicina Respiratoria, Córdoba
  - Sanatorio Allende Cerro, Córdoba
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Eastern Health Box Hill Hospital, Box Hill, Victoria
  - Monash Health-Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Institute for Respiratory Health - Midland, Midland, Western Australia
  - Institute for Respiratory Health, Nedlands, Western Australia
- Belgium (6):
  - AZORG, Aalst
  - ZAS Middelheim, Antwerp
  - CUB Hopital Erasmde, Brussels
  - Cliniques Universitaires St.-Luc, Brussels
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- Canada (5):
  - St.Paul's Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement Limited, Ajax, Ontario
  - St.Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - CIC Mauricie inc., Québec, Quebec
- Chile (6):
  - Centro de Investigacion Curico, Curicó, Maule Region
  - Centro Respiratorio Integral LTDA. (CENRESIN), Quillota, Región de Valparaíso
  - Centro de Investigación de Enfermedades Respiratorias e Inmunológicas (CIERI), Viña del Mar, Región de Valparaíso
  - CEC Centro Estudios Clinicos, Santiago, Santiago Metropolitan
  - Fundacion Medica San Cristobal, Santiago, Santiago Metropolitan
  - Biocinetic Ltda., Santiago, Santiago Metropolitan
- France (6):
  - Hôpital Avicennes, Bobigny
  - Hospices civils de Lyon - Hôpital Louis Pradel, Bron
  - CHU Caen Normandie, Caen
  - Assistance Publique Hôpitaux de Marseille - centre Hospitalier Régional de Marseille, Marseille
  - Rouen University Hospital, Rouen
  - Centre Hospitalier Régional Universitaire de Tours, Tours
- Germany (6):
  - RoMed Klinikum Rosenheim-Ellmaierstr. 23, Rosenheim, Bavaria
  - Zentralklinik Bad Berka GmbH Klinik für Pneumologie, Zentrum für Schlaf-und Beatmungsmedizin, Bad Berka
  - Prufstelle der GWT am Fachkrankenhaus Coswig, Coswig
  - uhrlandklinik Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - SLK Kliniken Heilbronn GmbH, Löwenstein
  - LMU Klinikum Medizinische Klinik und Poliklinik V, München
- Israel (9):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Rabin Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - The Hadassah University Medical Center Ein Kerem Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco" Presidio Ospedaliero Gaspare Rodolico, Catania
  - Azienda Unita Sanitaria Locale Della Romagna Ospedale "Gian Battista Morgagni - Luigi Pierantoni" di Forlì, Forlì
  - Azienda Ospedaliero-Universitaria di Modena Policlinico di Modena, Modena
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliero-Universitaria Senese, Siena
- New Zealand (2):
  - Canterbury Respiratory Research Group, Christchurch, Canterbury
  - Aotearoa Clinical Trials Trust- Middlemore Hospital, Auckland
- Peru (6):
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Clinica Internacional - Sede Lima, Lima
  - Unidad de Investigacion de Enfermedades Respiratorias- Clinica San Pablo -Surco, Lima
  - Clinica Ricardo Palma, Lima
  - Hospital Central de la Fuerza Aerea del Peru, Lima
  - Centro de Investigacion de Enfermedades Respiratorias - Clinica Providencia, Lima
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Papworth Hospital, Cambridge
  - NHS Lothian, Royal INfirmary of Edingburgh, Edinburgh
  - Guy's Hospital, London
  - Manchester University NHS Foundation Trust, North Manchester General Hospital, Manchester
  - NHS Tayside, Perth Royal Infirmary, Perth